CLINICAL TRIAL: NCT02595853
Title: A Novel Hemostatic Powder for the Endoscopic Treatment of Gastrointestinal Bleeding: Evaluation of Efficacy, Feasibility and Rebleeding Predictive Factors Results From a Multicenter Prospective Study Performed in Routine Practice
Brief Title: Efficacy of a Novel Hemostatic Powder in GI Bleeding
Acronym: GRAPHE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0077
Record Dates: First submitted 2015-10-29; First posted 2015-11-04 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Bleeding
Keywords: Upper GastroIntestinal bleeding, endoscopy, Hemospray
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study — All upper gastro-intestinal bleeding need endoscopic hemostasis. Endoscopic hemostasis conventional methods are injection of saline with epinephrine, placement of hemoclips and thermic or plasma coagulation. Hemospray™ will be sprayed onto bleeding lesions seen in endoscopy after failure of conventional methods or in salvage therapy at the discretion of endoscopists. Retrospective analysis of prospectively cellected data.

SUMMARY:
Hemospray™ is a new endoscopic hemostatic powder. Aims of this multicenter prospective study is to determine effectiveness of Hemospray™ on short and medium term in different clinical situations, predictive factors of rebleeding after Hemospray™ application, and feasibility of the application of hemostatic powder in routine clinical practice studying in a large sample of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over who need the use of Hemospray® under their care in an emergency.
* Upper gastrointestinal hemorrhage.
* Patients who received the information note of the study and agreeing to participate (non-oral opposition gathered in the patient's medical record)

Non Inclusion Criteria:

* Patient under guardianship, curatorship.
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who received hemostatic powder for upper GI bleeding will be included in the study. Pregnant and adult under guardianship will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of immediate cessation of bleeding observed in first-line per procedure or after failure of normal hemostasis techniques. | 30 days
  Percentage of immediate cessation of bleeding observed in first-line per procedure or after failure of normal hemostasis techniques.

SECONDARY OUTCOMES:
Rebleeding rate at days 8 and 30, defined as the percentage of patients with >2g/dL hemoglobin AND/OR exteriorization of hematemesis AND/OR exteriorization of melena | 30 days
  Rebleeding rate at days 8 and 30, defined as the percentage of patients with >2g/dL hemoglobin AND/OR exteriorization of hematemesis AND/OR exteriorization of melena

CONTACTS AND LOCATIONS:
Locations (19):
- France (18):
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Bordeuax University Hospital, Bordeaux
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - La Conception University Hospital, Marseille
  - La Timone University Hospital, Marseille
  - Nantes University Hospital, Nantes
  - Nîmes University Hospital, Nîmes
  - Cochin University Hospital, Paris
  - Georges Pompidou University Hospital (AP-HP), Paris
  - Henri Mondor University Hospital (AP-HP), Paris
  - Lariboisière University Hospital (AP-HP), Paris
  - Rouen University Hospital, Rouen
  - Saint-Brieuc University Hospital, Saint-Brieuc
  - Clinique des Cèdres, Toulouse
  - Tours University Hospital, Tours
  - Vichy Hospital, Vichy
- Monaco University Hospital, Monaco, Monaco

REFERENCES:
- [Derived] Haddara S, Jacques J, Lecleire S, Branche J, Leblanc S, Le Baleur Y, Privat J, Heyries L, Bichard P, Granval P, Chaput U, Koch S, Levy J, Godart B, Charachon A, Bourgaux JF, Metivier-Cesbron E, Chabrun E, Quentin V, Perrot B, Vanbiervliet G, Coron E. A novel hemostatic powder for upper gastrointestinal bleeding: a multicenter study (the "GRAPHE" registry). Endoscopy. 2016 Dec;48(12):1084-1095. doi: 10.1055/s-0042-116148. Epub 2016 Oct 19. PMID 27760437
- See also: Related Info — http://www.fmcgastro.org/textes-postus/postu-junior-2014/lendoscopie-a-luegw-2014/